CLINICAL TRIAL: NCT00523991
Title: A 24 Week, Randomized, Double-blind, Placebo Controlled, Multicenter Study to Evaluate the Efficacy and Safety of 18 MCG of Tiotropium Inhalation Capsules Administered by HandiHaler Once-daily Plus PRN Albuterol (Salbutamol) vs. Placebo Plus PRN Albuterol (Salbutamol) in Chronic Obstructive Pulmonary Disease Subjects Naive to Maintenance Therapy
Brief Title: Trial Comparing Tiotropium Inhalation Capsules vs Placebo in Chronic Obstructive Pulmonary Disease (COPD).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.365; A4471008 (Other: OTHER); 2006-006276-38 (EudraCT Number: EudraCT); NCT00460772 (obsolete NCT alias)
Record Dates: First submitted 2007-07-09; First posted 2007-09-03 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (2):
- placebo (Placebo Comparator): Oral inhalation once daily of placebo matching tiotropium via handihaler
  Interventions: Drug: Placebo
- tiotropium (Experimental): Oral inhalation once daily of 18mcg tiotropium via handihaler
  Interventions: Drug: tiotropium

INTERVENTIONS:
Drug: tiotropium — Oral inhalation once daily of 18mcg tiotropium via handihaler
  Arms: tiotropium
Drug: Placebo — Oral inhalation once daily of placebo matching tiotropium via handihaler
  Arms: placebo

SUMMARY:
A 24 week, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of 18mcg of tiotropium inhalation capsules administered by Handihaler once daily plus Pro Re Nata (PRN) albuterol (salbutamol) vs. placebo plus PRN albuterol (salbutamol) in chronic obstructive pulmonary disease subjects naive to maintenance therapy.

ELIGIBILITY:
Inclusion criteria:

All subjects must have a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) according to Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) guideline criteria:

post-bronchodilator Forced Expiratory Volume in one Second/Forced Vital Capacity (FEV1/FVC) ratio < 70% (visit 1).

Subjects must be GOLD Stage II and have a post-bronchodilator FEV1 >50% and < 80% of predicted normal (visit 1). Subjects must be current or ex-smokers with a smoking history of >=10 pack years.

Subjects must have a Medical Research Council (MRC) dyspnea score >= 2.

Exclusion criteria:

Subjects who have been treated with maintenance medications for chronic respiratory disease within six months prior to screening.

Subjects with significant diseases other than COPD. Subjects on chronic systemic corticosteroids.

Subjects with any upper and/or lower respiratory tract infection or COPD exacerbation in the 6 weeks prior to the initial visit 1 or during the screening period prior to visit 3 Subjects with a recent (past 6 months) myocardial infarction, any unstable or life threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year; or who have been hospitalized for cardiac failure during the past year.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2007-04; Primary Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (62):
- United States (17):
  - 205.365.1003 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.365.1004 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.365.1098 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 205.365.1023 Boehringer Ingelheim Investigational Site, Palo Alto, California
  - 205.365.1125 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.365.1024 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 205.365.1012 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.365.1086 Boehringer Ingelheim Investigational Site, Bloomington, Minnesota
  - 205.365.1006 Boehringer Ingelheim Investigational Site, Rochester, Minnesota
  - 205.365.1085 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 205.365.1010 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 205.365.1007 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 205.365.1080 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 205.365.1118 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.365.1033 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 205.365.1092 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 205.365.1122 Boehringer Ingelheim Investigational Site, Clarksburg, West Virginia
- Belgium (4):
  - 205.365.1103 Boehringer Ingelheim Investigational Site, Gilly
  - 205.365.1059 Boehringer Ingelheim Investigational Site, Leuven
  - 205.365.1057 Boehringer Ingelheim Investigational Site, Menen
  - 205.365.1058 Boehringer Ingelheim Investigational Site, Yvoir
- Canada (4):
  - 205.365.1042 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 205.365.1056 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 205.365.1104 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 205.365.1041 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
- Czechia (12):
  - 205.365.1064 Boehringer Ingelheim Investigational Site, Cvikov
  - 205.365.1107 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 205.365.1061 Boehringer Ingelheim Investigational Site, Karlovy Vary
  - 205.365.1077 Boehringer Ingelheim Investigational Site, Liberec
  - 205.365.1079 Boehringer Ingelheim Investigational Site, Neratovice
  - 205.365.1116 Boehringer Ingelheim Investigational Site, Pardubice
  - 205.365.1062 Boehringer Ingelheim Investigational Site, Prague
  - 205.365.1083 Boehringer Ingelheim Investigational Site, Prague
  - 205.365.1117 Boehringer Ingelheim Investigational Site, Prague
  - 205.365.1075 Boehringer Ingelheim Investigational Site, Strakonice
  - 205.365.1063 Boehringer Ingelheim Investigational Site, Tábor
  - 205.365.1076 Boehringer Ingelheim Investigational Site, Ústí nad Labem
- Germany (5):
  - 205.365.1055 Boehringer Ingelheim Investigational Site, Berlin
  - 205.365.1066 Boehringer Ingelheim Investigational Site, Berlin
  - 205.365.1054 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 205.365.1052 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 205.365.1050 Boehringer Ingelheim Investigational Site, Ulm
- Greece (3):
  - 205.365.1067 Boehringer Ingelheim Investigational Site, Athens
  - 205.365.1127 Boehringer Ingelheim Investigational Site, Athens
  - 205.365.1126 Boehringer Ingelheim Investigational Site, Thessaloniki
- Netherlands (4):
  - 205.365.1070 Boehringer Ingelheim Investigational Site, Enschede
  - 205.365.1072 Boehringer Ingelheim Investigational Site, Etten-Leur
  - 205.365.1071 Boehringer Ingelheim Investigational Site, Spijkenisse
  - 205.365.1069 Boehringer Ingelheim Investigational Site, Zutphen
- Portugal (3):
  - 205.365.1025 Boehringer Ingelheim Investigational Site, Amadora
  - 205.365.1020 Boehringer Ingelheim Investigational Site, Coimbra
  - 205.365.1022 Boehringer Ingelheim Investigational Site, Lisbon
- Ukraine (7):
  - 205.365.1128 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.365.1108 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.365.1110 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.365.1112 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.365.1114 Boehringer Ingelheim Investigational Site, Kiev
  - 205.365.1115 Boehringer Ingelheim Investigational Site, Kiev
  - 205.365.1113 Boehringer Ingelheim Investigational Site, Simferopol
- United Kingdom (3):
  - 205.365.44002 Boehringer Ingelheim Investigational Site, Garston, Watford
  - 205.365.44003 Boehringer Ingelheim Investigational Site, Harrow
  - 205.365.44004 Boehringer Ingelheim Investigational Site, Warminster

REFERENCES:
- [Derived] Troosters T, Sciurba FC, Decramer M, Siafakas NM, Klioze SS, Sutradhar SC, Weisman IM, Yunis C. Tiotropium in patients with moderate COPD naive to maintenance therapy: a randomised placebo-controlled trial. NPJ Prim Care Respir Med. 2014 May 20;24:14003. doi: 10.1038/npjpcrm.2014.3. PMID 24841833

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matching tiotropium via HandiHaler® + Pro Re Nata (PRN) albuterol
- Tiotropium: 18 mcg tiotropium via HandiHaler® + PRN albuterol
Period: Overall Study
Arm/Group | Placebo | Tiotropium
Started | 219 | 238
Completed | 198 | 211
Not Completed | 21 | 27
Not completed — Adverse Event | 6 | 5
Not completed — Protocol Violation | 1 | 4
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 7 | 17
Not completed — Other reason (not specified) | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo matching tiotropium via HandiHaler® + PRN albuterol
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium | Total
Number analyzed (Participants) | 219 | 238 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.6) | 61.2 (8.2) | 61.7 (8.4)
Age, Customized [Number; unit: participants]
  18-44 years | 8 | 7 | 15
  45-64 years | 121 | 151 | 272
  >=65 years | 90 | 80 | 170
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 72 | 144
  Male | 147 | 166 | 313
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 6 | 4 | 10
  White | 213 | 234 | 447

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lung Function as Measured by the Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve From 0-3h (AUC0-3h)
Description: Change = Week 24 Value - Baseline Value
Time Frame: baseline, week 24
Population: Full Analysis Set (FAS): All randomized subjects who received at least 1 dose of study drug, had baseline and at least 1 post baseline data measurement available for the primary endpoint
Measure: Least Squares Mean (Standard Error); unit: litres * hours
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres * hours | -0.06 (0.02) | 0.16 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Test type: Superiority or Other; p < 0.001, ANCOVA — There was only one primary endpoint and the p-value was not adjusted for multiple comparisons. Mean Difference (Final Values) means difference in LS-Means; The analysis of covariance model included treatment, site, and trough forced expiratory volume in 1 second at baseline in the model; Mean Difference (Final Values) = 0.23, 95% CI [0.18 to 0.27]

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1)(Baseline)
Description: Trough FEV1 defined as the FEV1 measured at 10 minutes prior to the end of the dosing interval, approximately 24 hours post drug administration. Baseline FEV1 was the pre-treatment FEV1 measured at Week 0 in the morning 10 minutes prior to the administration of the first dose of the study medication.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.71 (0.45) | 1.74 (0.46)

3. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (at Week 8)
Description: as for outcome 2
Time Frame: Baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.03 (0.21) | 0.12 (0.21)

4. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (at Week 16)
Description: as for outcome 2
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.06 (0.21) | 0.09 (0.27)

5. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (at Week 24)
Description: as for outcome 2
Time Frame: Baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.08 (0.02) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — All secondary analyses are exploratory and therefore no corrections for multiple hypotheses testing are made. The results have to be interpreted in a descriptive manner; Terms include treatment, site, and trough forced expiratory volume in 1 second at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.14, 95% CI [0.09 to 0.18]

6. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (Baseline)
Description: Peak FEV1 defined as the maximum of the observed values over 30, 60, 120, and 180 minutes post-dose for FEV1.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.71 (0.45) | 1.74 (0.46)

7. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 8)
Description: Peak FEV1 defined as the maximum of the observed values over 30, 60, 120, and 180 minutes post-dose for FEV1. Peak response was defined as the change from baseline to the peak FEV1 value at the final visit.
Time Frame: Baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.09 (0.22) | 0.31 (0.24)

8. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 16)
Description: as for outcome 7
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.05 (0.24) | 0.29 (0.28)

9. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 24)
Description: as for outcome 7
Time Frame: Baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.02 (0.02) | 0.26 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Terms include treatment, site, and peak forced expiratory volume in 1 second at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.24, 95% CI [0.19 to 0.29]

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (Baseline, Pre-dose)
Description: Forced expiratory volume in 1 second (baseline, pre-dose)
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.71 (0.45) | 1.74 (0.46)

11. Secondary Outcome: Forced Expiratory Volume in 1 Second (Baseline, 30 Minutes)
Description: Forced expiratory volume in 1 second (baseline, 30 minutes)
Time Frame: baseline, 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.73 (0.45) | 1.87 (0.47)

12. Secondary Outcome: Forced Expiratory Volume in 1 Second (Baseline, 60 Minutes)
Description: Forced expiratory volume in 1 second (baseline, 60 minutes)
Time Frame: baseline, 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.74 (0.47) | 1.90 (0.47)

13. Secondary Outcome: Forced Expiratory Volume in 1 Second (Baseline, 120 Minutes)
Description: Forced expiratory volume in 1 second (baseline, 120 minutes)
Time Frame: Baseline, 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.75 (0.48) | 1.92 (0.49)

14. Secondary Outcome: Forced Expiratory Volume in 1 Second (Baseline, 180 Minutes)
Description: Forced expiratory volume in 1 second (baseline, 180 minutes)
Time Frame: Baseline, 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 1.76 (0.48) | 1.94 (0.48)

15. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (at Week 8, Pre-dose)
Description: Change from baseline in forced expiratory volume in 1 second (at week 8, pre-dose)
Time Frame: baseline, week 8, pre-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.03 (0.21) | 0.12 (0.21)

16. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (at Week 8, 30 Minutes)
Description: Change from baseline in forced expiratory volume in 1 second (at week 8, 30 minutes)
Time Frame: Baseline, week 8, 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.00 (0.22) | 0.20 (0.22)

17. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (at Week 8, 60 Minutes)
Description: Change from baseline in forced expiratory volume in 1 second (at week 8, 60 minutes)
Time Frame: baseline, week 8, 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.01 (0.24) | 0.22 (0.24)

18. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (at Week 8, 120 Minutes)
Description: Change from baseline in forced expiratory volume in 1 second (at week 8, 120 minutes)
Time Frame: baseline, week 8, 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.01 (0.23) | 0.24 (0.23)

19. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (at Week 8, 180 Minutes)
Description: Change from baseline in forced expiratory volume in 1 second (at week 8, 180 minutes)
Time Frame: baseline, week 8, 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.01 (0.22) | 0.24 (0.25)

20. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (at Week 16, Pre-dose)
Description: Change from baseline in forced expiratory volume in 1 second (at week 16, pre-dose)
Time Frame: baseline, week 16, pre-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.06 (0.21) | 0.09 (0.27)

21. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 16, 30 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 16, 30 minutes)
Time Frame: Baseline, week 16, 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.02 (0.24) | 0.19 (0.27)

22. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 16, 60 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 16, 60 minutes)
Time Frame: baseline, week 16, 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.02 (0.24) | 0.21 (0.27)

23. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 16, 120 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 16, 120 minutes)
Time Frame: baseline, week 16, 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.03 (0.24) | 0.22 (0.28)

24. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 16, 180 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 16, 180 minutes)
Time Frame: baseline, week 16, 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.02 (0.24) | 0.22 (0.28)

25. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 24, Pre-dose)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 24, pre-dose)
Time Frame: baseline, week 24, pre-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.08 (0.02) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Terms include treatment, site, and forced expiratory volume in 1 second at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.14, 95% CI [0.09 to 0.18]

26. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 24, 30 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 24, 30 minutes)
Time Frame: baseline, week 24, 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.05 (0.02) | 0.15 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI [0.16 to 0.25]

27. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 24, 60 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 24, 60 minutes)
Time Frame: baseline, week 24, 60 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.05 (0.02) | 0.18 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium vesus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI [0.18 to 0.28]

28. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 24, 120 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 24, 120 minutes)
Time Frame: baseline, week 24, 120 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.06 (0.02) | 0.18 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI [0.20 to 0.29]

29. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (at Week 24, 180 Minutes)
Description: Change from baseline in peak forced expiratory volume in 1 second (at week 24, 180 minutes)
Time Frame: baseline, week 24, 180 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.05 (0.02) | 0.20 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.25, 95% CI [0.20 to 0.30]

30. Secondary Outcome: FVC AUC0-3 at Baseline
Description: Forced vital capacity (FVC) area under the curve from 0-3 hours (AUC0-3h)
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres * hours
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres * hours | 3.17 (0.82) | 3.24 (0.81)

31. Secondary Outcome: FVC AUC0-3 at Week 8 Minus Baseline
Description: Change from baseline in Forced vital capacity (FVC) area under the curve from 0-3 hours (AUC0-3h) (week 8)
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres * hours
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres * hours | -0.01 (0.35) | 0.28 (0.39)

32. Secondary Outcome: FVC AUC0-3 at Week 16 Minus Baseline
Description: Change from baseline in Forced vital capacity (FVC) area under the curve from 0-3 hours (AUC0-3h)(week 16)
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres * hours
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres * hours | -0.06 (0.39) | 0.24 (0.43)

33. Secondary Outcome: FVC AUC0-3 at Week 24 Minus Baseline
Description: Change from baseline in Forced vital capacity (FVC) area under the curve from 0-3 hours (AUC0-3h) (week 24)
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres * hours
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres * hours | -0.11 (0.03) | 0.19 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms include treatment, site, and forced vital capacity area under the curve at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.31, 95% CI [0.24 to 0.38]

34. Secondary Outcome: Trough Forced Vital Capacity (Baseline)
Description: Trough FVC defined as the FVC measured at 10 minutes prior to the end of the dosing interval, approximately 24 hours post drug administration. Baseline FVC was the pre-treatment FVC measured at Week 0 in the morning 10 minutes prior to the administration of the first dose of the study medication.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.17 (0.82) | 3.24 (0.81)

35. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (at Week 8)
Description: as for outcome 34
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.06 (0.33) | 0.16 (0.38)

36. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (at Week 16)
Description: as for outcome 34
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.13 (0.37) | 0.10 (0.42)

37. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (at Week 24)
Description: as for outcome 34
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.14 (0.03) | 0.07 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms include treatment, site, and trough forced vital capacity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.21, 95% CI [0.14 to 0.28]

38. Secondary Outcome: Peak Forced Vital Capacity (FVC) (Baseline)
Description: Peak FEV1 defined as the maximum of the observed values over 30, 60, 120, and 180 minutes post-dose for FEV1.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.17 (0.82) | 3.24 (0.81)

39. Secondary Outcome: Change From Baseline in Peak Forced Vital Capacity (at Week 8)
Description: as for outcome 7
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.13 (0.34) | 0.43 (0.40)

40. Secondary Outcome: Change From Baseline in Peak Forced Vital Capacity (at Week 16)
Description: as for outcome 7
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.08 (0.40) | 0.38 (0.44)

41. Secondary Outcome: Change From Baseline in Peak Forced Vital Capacity (at Week 24)
Description: as for outcome 7
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.06 (0.04) | 0.40 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms include treatment, site, and peak forced vital capacity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.33, 95% CI [0.24 to 0.42]

42. Secondary Outcome: Forced Vital Capacity (Baseline, Pre-dose)
Description: Forced vital capacity (baseline, pre-dose)
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.17 (0.82) | 3.24 (0.81)

43. Secondary Outcome: Forced Vital Capacity (Baseline, 30 Minutes)
Description: Forced vital capacity (baseline, 30 minutes)
Time Frame: baseline, 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.20 (0.82) | 3.45 (0.83)

44. Secondary Outcome: Forced Vital Capacity (Baseline, 60 Minutes)
Description: Forced vital capacity (baseline, 60 minutes)
Time Frame: baseline, 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.22 (0.85) | 3.48 (0.84)

45. Secondary Outcome: Forced Vital Capacity (Baseline, 120 Minutes)
Description: Forced vital capacity (baseline, 120 minutes)
Time Frame: baseline, 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.21 (0.86) | 3.49 (0.85)

46. Secondary Outcome: Forced Vital Capacity (Baseline, 180 Minutes)
Description: Forced vital capacity (baseline, 180 minutes)
Time Frame: baseline, 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 3.21 (0.83) | 3.50 (0.85)

47. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 8, Pre-dose)
Description: Change from baseline in forced vital capacity (week 8, pre-dose)
Time Frame: baseline, week 8, pre-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.06 (0.33) | 0.16 (0.38)

48. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 8, 30 Minutes)
Description: Change from baseline in forced vital capacity (week 8, 30 minutes)
Time Frame: baseline, week 8, 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.00 (0.35) | 0.27 (0.40)

49. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 8, 60 Minutes)
Description: Change from baseline in forced vital capacity (week 8, 60 minutes)
Time Frame: baseline, week 8, 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.00 (0.37) | 0.29 (0.43)

50. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 8, 120 Minutes)
Description: Change from baseline in forced vital capacity (week 8, 120 minutes)
Time Frame: baseline, week 8, 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.02 (0.39) | 0.30 (0.40)

51. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 8, 180 Minutes)
Description: Change from baseline in forced vital capacity (week 8, 180 minutes)
Time Frame: baseline, week 8, 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | 0.00 (0.37) | 0.30 (0.43)

52. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 16, Pre-dose)
Description: Change from baseline in forced vital capacity (week 16, pre-dose)
Time Frame: baseline, week 16, pre-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.13 (0.37) | 0.10 (0.42)

53. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 16, 30 Minutes)
Description: Change from baseline in forced vital capacity (week 16, 30 minutes)
Time Frame: baseline, week 16, 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.06 (0.39) | 0.24 (0.45)

54. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 16, 60 Minutes)
Description: Change from baseline in forced vital capacity (week 16, 60 minutes)
Time Frame: baseline, week 16, 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.05 (0.41) | 0.27 (0.45)

55. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 16, 120 Minutes)
Description: Change from baseline in forced vital capacity (week 16, 120 minutes)
Time Frame: baseline, week 16, 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.05 (0.41) | 0.26 (0.45)

56. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 16, 180 Minutes)
Description: Change from baseline in forced vital capacity (week 16, 180 minutes)
Time Frame: baseline, week 16, 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.05 (0.42) | 0.26 (0.45)

57. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 24, Pre-dose)
Description: Change from baseline in forced vital capacity (week 24, pre-dose)
Time Frame: baseline, week 24, pre-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.14 (0.03) | 0.07 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms include treatment, site, and forced vital capacity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.21, 95% CI [0.14 to 0.28]

58. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 24, 30 Minutes)
Description: Change from baseline in forced vital capacity (week 24, 30 minutes)
Time Frame: baseline, week 24, 30 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.10 (0.03) | 0.19 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 57, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI [0.21 to 0.36]

59. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 24, 60 Minutes)
Description: Change from baseline in forced vital capacity (week 24, 60 minutes)
Time Frame: baseline, week 24, 60 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.07 (0.03) | 0.23 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 57, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI [0.23 to 0.38]

60. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 24, 120 Minutes)
Description: Change from baseline in forced vital capacity (week 24, 120 minutes)
Time Frame: baseline, week 24, 120 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.11 (0.03) | 0.22 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 57, analysis 1]; Mean Difference (Final Values) = 0.33, 95% CI [0.25 to 0.40]

61. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Week 24, 180 Minutes)
Description: Change from baseline in forced vital capacity (week 24, 180 minutes)
Time Frame: baseline, week 24, 180 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
litres | -0.07 (0.04) | 0.29 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 57, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI [0.26 to 0.45]

62. Secondary Outcome: Albuterol Use p.r.n. (Baseline)
Description: Number of days that participants used albuterol prn per week
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
days | 2.1 (2.76) | 1.8 (2.63)

63. Secondary Outcome: Change From Baseline in Albuterol Use p.r.n. - (Week 4)
Description: Difference in number of days that participants used albuterol prn per week between week 4 and baseline
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
days | -0.2 (1.71) | -0.2 (2.07)

64. Secondary Outcome: Change From Baseline in Albuterol Use p.r.n. - (Week 8)
Description: Difference in number of days that participants used albuterol prn per week between week 8 and baseline
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 225
days | -0.3 (2.13) | -0.3 (1.96)

65. Secondary Outcome: Change From Baseline in Albuterol Use p.r.n. -(Week 12)
Description: Difference in number of days that participants used albuterol prn per week between week 12 and baseline
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 206 | 220
days | -0.3 (2.16) | -0.3 (2.09)

66. Secondary Outcome: Change From Baseline in Albuterol Use p.r.n. - (Week 16)
Description: Difference in number of days that participants used albuterol prn per week between week 16 and baseline
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 203 | 215
days | -0.4 (2.10) | -0.3 (2.26)

67. Secondary Outcome: Change From Baseline in Albuterol Use p.r.n. -(Week 20)
Description: Difference in number of days that participants used albuterol prn per week between week 20 and baseline
Time Frame: baseline, week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 201 | 212
days | -0.4 (2.34) | -0.3 (2.21)

68. Secondary Outcome: Change From Baseline in Albuterol Use p.r.n. - (Week 24)
Description: Difference in number of days that participants used albuterol prn per week between week 24 and baseline
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 201 | 216
days | -0.64 (0.18) | -0.62 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.927, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms include treatment, site, and albuterol use at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.02, 95% CI [-0.38 to 0.41]

69. Secondary Outcome: Number of Participants With Categorical Scores on Physician's Global Assessment (Baseline)
Description: The physician's global assessment reflected the physician's opinion of the participant's overall clinical condition with respect to COPD. The evaluation was based on the participant's use of concomitant medications, as well as the number and severity of COPD exacerbations and related emergency room visits and/or hospitalizations since the last visit. The frequency and severity of symptoms ( cough, dyspnea, wheezing) and the impact of these on the participant's ability to exercise were considered.
  Range: 1-2 = Poor, 3-4 = Fair 5-6 = Good, 7-8 = Excellent.
Time Frame: baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 207 | 227
Participants
  Poor/Fair | 62 | 78
  Good | 122 | 132
  Excellent | 23 | 17
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.174, Cochran-Mantel-Haenszel; Site as stratum

70. Secondary Outcome: Number of Participants With Categorical Scores on Physician's Global Assessment (Week 12)
Description: as for outcome 69
Time Frame: week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 204 | 220
Participants
  Poor/Fair | 49 | 50
  Good | 135 | 134
  Excellent | 20 | 36
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.186, Cochran-Mantel-Haenszel; Site as stratum

71. Secondary Outcome: Number of Participants With Categorical Scores on Physician's Global Assessment (Week 24)
Description: as for outcome 69
Time Frame: week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 201 | 216
Participants
  Poor/Fair | 51 | 41
  Good | 128 | 136
  Excellent | 22 | 39
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.045, Cochran-Mantel-Haenszel; Site as stratum

72. Secondary Outcome: Number of Participants With Categorical Scores on Patient's Global Assessment (Baseline)
Description: The patient's global assessment was based on the subject's need to take additional medications for breathing, their need for emergency room or hospital visits for COPD, and severity and amount of coughing, wheezing, and/or breathing discomfort experienced, and the impact of these symptoms on the subject's ability to exercise and perform daily activities.
  Range: 1-2 = Poor, 3-4 = Fair 5-6 = Good, 7-8 = Excellent.
Time Frame: baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 206 | 227
Participants
  Poor/Fair | 72 | 95
  Good | 111 | 117
  Excellent | 23 | 15
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.223, Cochran-Mantel-Haenszel; Site as stratum

73. Secondary Outcome: Number of Participants With Categorical Scores on Patient's Global Assessment (Week 12)
Description: as for outcome 72
Time Frame: week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 206 | 220
Participants
  Poor/Fair | 62 | 53
  Good | 127 | 132
  Excellent | 17 | 35
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel; Site as stratum

74. Secondary Outcome: Number of Participants With Categorical Scores on Patient's Global Assessment (Week 24)
Description: as for outcome 72
Time Frame: week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 201 | 216
Participants
  Poor/Fair | 66 | 56
  Good | 116 | 128
  Excellent | 19 | 32
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel; Site as stratum

75. Secondary Outcome: Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Baseline)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment.
  Absenteeism, Presenteeism, Work productivity loss, Activity Impairment Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 206 | 227
units on a scale | 25.4 (21.43) | 28 (22.32)

76. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Week 4)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment. Difference refers to change in scale between week 4 and baseline.
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 205 | 225
units on a scale | 0.34 (1.64) | 0.98 (1.53)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.729, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LS Means; Mean Difference (Final Values) = 0.64, 95% CI [-2.97 to 4.24]

77. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Week 8)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment. Difference refers to change in scale between week 8 and baseline.
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 206 | 225
units on a scale | 2.12 (1.54) | -0.38 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.149, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 76, analysis 1]; Mean Difference (Final Values) = -2.50, 95% CI [-5.90 to 0.90]

78. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Week 12)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment. Difference refers to change in scale between week 12 and baseline.
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 205 | 217
units on a scale | -0.54 (1.58) | -1.07 (1.51)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.763, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.53, 95% CI [-4.00 to 2.93]

79. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Week 16)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment. Difference refers to change in scale between week 16 and baseline.
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 200 | 214
units on a scale | 4.47 (1.64) | 2.62 (1.54)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.313, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 76, analysis 1]; Mean Difference (Final Values) = -1.85, 95% CI [-5.45 to 1.75]

80. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Week 20)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment. Difference refers to change in scale between week 20 and baseline.
Time Frame: baseline, week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 200 | 211
units on a scale | 4.32 (1.62) | 3.52 (1.70)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.682, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 76, analysis 1]; Mean Difference (Final Values) = -0.79, 95% CI [-4.60 to 3.01]

81. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment Due to Health (Week 24)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment. Scores range from 0 to 100 for each of the above 4 types; higher scores indicate greater impairment. Difference refers to change in scale between week 24 and baseline.
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 198 | 215
units on a scale | 5.26 (1.64) | 1.51 (1.54)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.043, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 76, analysis 1]; Mean Difference (Final Values) = -3.76, 95% CI [-7.39 to -0.13]

82. Secondary Outcome: Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health
Description: as for outcome 75
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 75 | 89
units on a scale | 17.2 (20.24) | 21.1 (21.08)

83. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health (Week 4)
Description: as for outcome 76
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 69 | 83
units on a scale | -2.03 (2.21) | -2.64 (2.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.823, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.61, 95% CI [-6.01 to 4.79]

84. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health (Week 8)
Description: as for outcome 77
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 68 | 77
units on a scale | 0.41 (2.71) | -0.61 (2.60)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.767, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -1.03, 95% CI [-7.86 to 5.81]

85. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health (Week 12)
Description: as for outcome 78
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 68 | 76
units on a scale | -0.32 (1.91) | 0.46 (1.84)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.754, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.77, 95% CI [-4.12 to 5.67]

86. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health (Week 16)
Description: as for outcome 79
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 67 | 74
units on a scale | 3.68 (2.46) | 3.66 (2.33)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.995, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.02, 95% CI [-6.31 to 6.27]

87. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health (Week 20)
Description: as for outcome 80
Time Frame: baseline, week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 66 | 73
units on a scale | 4.27 (2.55) | 3.08 (2.44)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.720, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -1.19, 95% CI [-7.77 to 5.39]

88. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Impairment While Working Due to Health (Week 24)
Description: as for outcome 81
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 64 | 71
units on a scale | 4.04 (2.43) | -1.84 (2.29)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.064, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 76, analysis 1]; Mean Difference (Final Values) = -5.88, 95% CI [-12.10 to 0.35]

89. Secondary Outcome: Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Baseline)
Description: as for outcome 75
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 74 | 89
units on a scale | 19.3 (22.17) | 22.0 (22.06)

90. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Week 4)
Description: as for outcome 76
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 69 | 83
units on a scale | -2.39 (2.48) | -3.50 (2.31)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.718, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -1.11, 95% CI [-7.21 to 4.98]

91. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Week 8)
Description: as for outcome 77
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 68 | 77
units on a scale | -0.62 (2.96) | -1.04 (2.86)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.912, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.42, 95% CI [-7.90 to 7.06]

92. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Week 12)
Description: as for outcome 78
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 68 | 76
units on a scale | 0.32 (2.09) | 4.11 (2.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.162, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 3.79, 95% CI [-1.55 to 9.13]

93. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Week 16)
Description: as for outcome 79
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 67 | 74
units on a scale | 2.20 (2.78) | 4.79 (2.64)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.471, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 2.59, 95% CI [-4.51 to 9.69]

94. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Week 20)
Description: as for outcome 80
Time Frame: baseline, week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 66 | 73
units on a scale | 3.93 (2.58) | 4.10 (2.50)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.961, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.16, 95% CI [-6.52 to 6.84]

95. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Overall Work Impairment Due to Health (Week 24)
Description: as for outcome 81
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 63 | 71
units on a scale | 2.20 (2.70) | -2.70 (2.50)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.158, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -4.90, 95% CI [-11.73 to 1.94]

96. Secondary Outcome: Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Baseline)
Description: as for outcome 75
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 76 | 94
units on a scale | 5.5 (19.31) | 2.7 (12.35)

97. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Week 4)
Description: as for outcome 76
Time Frame: baseline, week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 71 | 88
units on a scale | -1.89 (1.96) | -0.15 (1.77)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.469, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 1.74, 95% CI [-3.01 to 6.49]

98. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Week 8)
Description: as for outcome 77
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 71 | 84
units on a scale | -1.94 (2.62) | 3.85 (2.43)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.079, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 5.79, 95% CI [-0.68 to 12.26]

99. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Week 12)
Description: as for outcome 78
Time Frame: baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 71 | 80
units on a scale | 0.12 (1.63) | 4.22 (1.55)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 4.10, 95% CI [-0.02 to 8.23]

100. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Week 16)
Description: as for outcome 79
Time Frame: baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 71 | 80
units on a scale | -3.39 (1.49) | 0.04 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.075, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 3.43, 95% CI [-0.35 to 7.21]

101. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Week 20)
Description: as for outcome 80
Time Frame: baseline, week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 69 | 78
units on a scale | 0.51 (1.13) | 2.00 (1.08)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.306, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 1.50, 95% CI [-1.39 to 4.38]

102. Secondary Outcome: Change From Baseline in Work Productivity as Assessed by the Work Productivity and Activity Impairment (WPAI) Questionnaire: Work Time Missed Due to Health (Week 24)
Description: as for outcome 81
Time Frame: baseline, week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 68 | 76
units on a scale | 0.96 (2.00) | -1.37 (1.86)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.363, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and work productivity at baseline Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -2.33, 95% CI [-7.39 to 2.73]

103. Secondary Outcome: Physical Activity (Light Intensity; Baseline) in Logarithm of Average Time Spent in Minutes Per Day
Description: Light intensity is less than three metabolic equivalents.
  Metabolic equivalent threshold (MET): Unit used to estimate the metabolic cost of physical activity, in terms of multiples of the subject's resting metabolic rate. One metabolic equivalent is, by convention, 3.5 ml of O2 uptake per minute per kilogram body weight, and theoretically approximates the resting metabolic rate.
  ln in measure value unit means natural logarithm.
Time Frame: baseline
Population: Activity evaluable set population: All subjects included in the Full Analysis Set (FAS), who had physical activity and energy expenditure data available for >= 12 weeks, and who wore the activity monitor for >11 hours for at least 4 days
Measure: Mean (Standard Deviation); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 184 | 203
ln(minutes) | 6.9 (0.24) | 6.8 (0.27)

104. Secondary Outcome: Change From Baseline in Physical Activity (Light Intensity; Week 4) in Logarithm of Average Time Spent in Minutes Per Day
Description: Light intensity is less than three metabolic equivalents
  Metabolic equivalent threshold (MET): Unit used to estimate the metabolic cost of physical activity, in terms of multiples of the subject's resting metabolic rate. One metabolic equivalent is, by convention, 3.5 ml of O2 uptake per minute per kilogram body weight, and theoretically approximates the resting metabolic rate.
  ln in measure value unit means natural logarithm
Time Frame: baseline, week 4
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 188
ln(minutes) | 0.03 (0.01) | 0.02 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.668, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.01, 95% CI [-0.03 to 0.02]

105. Secondary Outcome: Change From Baseline in Physical Activity (Light Intensity; Week 8) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 104
Time Frame: baseline, week 8
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 184
ln(minutes) | 0.02 (0.01) | 0.03 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.780, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.00, 95% CI [-0.02 to 0.03]

106. Secondary Outcome: Change From Baseline in Physical Activity (Light Intensity; Week 12) in Logarithm of Average Time Spent in Minutes Per Day
Description: Light intensity defined as less than three metabolic equivalents.
  Metabolic equivalent threshold (MET): Unit used to estimate the metabolic cost of physical activity, in terms of multiples of the subject's resting metabolic rate. One metabolic equivalent is, by convention, 3.5 ml of O2 uptake per minute per kilogram body weight, and theoretically approximates the resting metabolic rate.
  ln in measure value unit means natural logarithm
Time Frame: baseline, week 12
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 173 | 185
ln(minutes) | 0.03 (0.01) | 0.02 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.610, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.01, 95% CI [-0.03 to 0.02]

107. Secondary Outcome: Change From Baseline in Physical Activity (Light Intensity; Week 16) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 104
Time Frame: baseline, week 16
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 171 | 183
ln(minutes) | 0.03 (0.01) | 0.04 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.554, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.01, 95% CI [-0.02 to 0.04]

108. Secondary Outcome: Change From Baseline in Physical Activity (Light Intensity; Week 20) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 104
Time Frame: baseline, week 20
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 172 | 182
ln(minutes) | 0.03 (0.01) | 0.04 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.549, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.01, 95% CI [-0.02 to 0.04]

109. Secondary Outcome: Change From Baseline in Physical Activity (Light Intensity; Week 24) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 104
Time Frame: baseline, week 24
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 167 | 186
ln(minutes) | 0.02 (0.02) | 0.03 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.568, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.01, 95% CI [-0.02 to 0.04]

110. Secondary Outcome: Physical Activity (Moderate or Higher Intensity; Baseline) in Logarithm of Average Time Spent in Minutes Per Day
Description: Moderate or higher intensity is greater than or equal to three metabolic equivalents
  Metabolic equivalent threshold (MET): Unit used to estimate the metabolic cost of physical activity, in terms of multiples of the subject's resting metabolic rate. One metabolic equivalent is, by convention, 3.5 ml of O2 uptake per minute per kilogram body weight, and theoretically approximates the resting metabolic rate.
  ln in measure value unit means natural logarithm
Time Frame: baseline
Population: as for outcome 103
Measure: Mean (Standard Deviation); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 184 | 203
ln(minutes) | 4.2 (0.96) | 4.3 (0.92)

111. Secondary Outcome: Change From Baseline in Physical Activity (Moderate or Higher Intensity; Week 4) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 110
Time Frame: baseline, week 4
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 174 | 187
ln(minutes) | -0.06 (0.06) | -0.12 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.358, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.06, 95% CI [-0.18 to 0.07]

112. Secondary Outcome: Change From Baseline in Physical Activity (Moderate or Higher Intensity; Week 8) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 110
Time Frame: baseline, week 8
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 184
ln(minutes) | 0.01 (0.05) | -0.06 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.219, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.08, 95% CI [-0.20 to 0.05]

113. Secondary Outcome: Change From Baseline in Physical Activity (Moderate or Higher Intensity; Week 12) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 110
Time Frame: baseline, week 12
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 173 | 183
ln(minutes) | -0.14 (0.07) | -0.09 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.518, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.05, 95% CI [-0.10 to 0.19]

114. Secondary Outcome: Change From Baseline in Physical Activity (Moderate or Higher Intensity; Week 16) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 110
Time Frame: baseline, week 16
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 171 | 183
ln(minutes) | -0.26 (0.07) | -0.20 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.455, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.06, 95% CI [-0.09 to 0.21]

115. Secondary Outcome: Change From Baseline in Physical Activity (Moderate or Higher Intensity; Week 20) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 110
Time Frame: baseline, week 20
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 172 | 182
ln(minutes) | -0.20 (0.07) | -0.20 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.927, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.01, 95% CI [-0.16 to 0.15]

116. Secondary Outcome: Change From Baseline in Physical Activity (Moderate or Higher Intensity; Week 24) in Logarithm of Average Time Spent in Minutes Per Day
Description: as for outcome 110
Time Frame: baseline, week 24
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: ln(minutes)
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 167 | 186
ln(minutes) | -0.19 (0.08) | -0.20 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.933, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and logarithm of baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.01, 95% CI [-0.17 to 0.16]

117. Secondary Outcome: Number of Participants With Healthy Lifestyle (Baseline)
Description: Healthy lifestyle defined as 30 minutes of activity > 3 metabolic equivalent levels for 70% of eligible days. Two categories: Yes, no
Time Frame: baseline
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 184 | 203
Participants
  Yes | 126 | 143
  No | 58 | 60
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.996, Cochran-Mantel-Haenszel; Site as stratum

118. Secondary Outcome: Number of Participants With Healthy Lifestyle (Week 4)
Description: as for outcome 117
Time Frame: week 4
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 187 | 204
Participants
  Yes | 129 | 154
  No | 58 | 50
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.196, Cochran-Mantel-Haenszel; Site as stratum

119. Secondary Outcome: Number of Participants With Healthy Lifestyle (Week 8)
Description: as for outcome 117
Time Frame: week 8
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 191 | 197
Participants
  Yes | 125 | 137
  No | 66 | 60
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.800, Cochran-Mantel-Haenszel; Site as stratum

120. Secondary Outcome: Number of Participants With Healthy Lifestyle (Week 12)
Description: as for outcome 117
Time Frame: week 12
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 189 | 199
Participants
  Yes | 118 | 139
  No | 71 | 60
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.215, Cochran-Mantel-Haenszel; Site as stratum

121. Secondary Outcome: Number of Participants With Healthy Lifestyle (Week 16)
Description: as for outcome 117
Time Frame: week 16
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 187 | 193
Participants
  Yes | 116 | 133
  No | 71 | 60
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.205, Cochran-Mantel-Haenszel; Site as stratum

122. Secondary Outcome: Number of Participants With Healthy Lifestyle (Week 20)
Description: as for outcome 117
Time Frame: week 20
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 188 | 190
Participants
  Yes | 127 | 134
  No | 61 | 56
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.622, Cochran-Mantel-Haenszel; Site as stratum

123. Secondary Outcome: Number of Participants With Healthy Lifestyle (Week 24)
Description: as for outcome 117
Time Frame: week 24
Population: as for outcome 103
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 182 | 196
Participants
  Yes | 118 | 136
  No | 64 | 60
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.446, Cochran-Mantel-Haenszel; Site as stratum

124. Secondary Outcome: Active Energy Expenditure (Baseline)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline
Population: as for outcome 103
Measure: Mean (Standard Deviation); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 184 | 203
kilo calories per day | 0.87 (0.46) | 0.87 (0.46)

125. Secondary Outcome: Change From Baseline in Active Energy Expenditure (Week 4)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline, week 4
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 188
kilo calories per day | -0.04 (0.03) | -0.03 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.819, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 0.01, 95% CI [-0.05 to 0.06]

126. Secondary Outcome: Change From Baseline in Active Energy Expenditure (Week 8)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline, week 8
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 184
kilo calories per day | 0.01 (0.03) | -0.03 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.204, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.04, 95% CI [-0.10 to 0.02]

127. Secondary Outcome: Change From Baseline in Active Energy Expenditure (Week 12)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline, week 12
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 173 | 185
kilo calories per day | -0.05 (0.03) | -0.06 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.670, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.01, 95% CI [-0.08 to 0.05]

128. Secondary Outcome: Change From Baseline in Active Energy Expenditure (Week 16)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline, week 16
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 171 | 183
kilo calories per day | -0.07 (0.03) | -0.09 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.630, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.02, 95% CI [-0.09 to 0.06]

129. Secondary Outcome: Change From Baseline in Active Energy Expenditure (Week 20)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline, week 20
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 172 | 182
kilo calories per day | -0.08 (0.04) | -0.09 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.704, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.02, 95% CI [-0.10 to 0.07]

130. Secondary Outcome: Change From Baseline in Active Energy Expenditure (Week 24)
Description: The amount of energy (kcal/day) that a person uses while physically active.
Time Frame: baseline, week 24
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: kilo calories per day
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 167 | 186
kilo calories per day | -0.08 (0.04) | -0.10 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.579, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -0.02, 95% CI [-0.11 to 0.06]

131. Secondary Outcome: Number of Steps Per Day (Baseline)
Description: Number of steps per day (baseline)
Time Frame: baseline
Population: as for outcome 103
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 184 | 203
Steps | 7343.4 (3711.8) | 7366.1 (3816.0)

132. Secondary Outcome: Change From Baseline in Number of Steps Per Day (Week 4)
Description: Change from baseline in number of steps per day (week 4)
Time Frame: baseline, week 4
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 188
Steps | -263.91 (203.37) | -287.45 (189.24)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.916, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -23.54, 95% CI [-464.02 to 416.94]

133. Secondary Outcome: Change From Baseline in Number of Steps Per Day(Week 8)
Description: Change from baseline in number of steps per day (week 8)
Time Frame: baseline, week 8
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 175 | 184
Steps | -121.66 (214.73) | -153.09 (203.84)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.899, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = -31.42, 95% CI [-520.19 to 457.34]

134. Secondary Outcome: Change From Baseline in Number of Steps Per Day (Week 12)
Description: Change from baseline in Number of steps per day (week 12)
Time Frame: baseline, week 12
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 173 | 185
Steps | -351.30 (239.39) | -169.31 (221.09)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; placebo versus tiotropium; Test type: Superiority or Other; p = 0.495, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 181.99, 95% CI [-341.75 to 705.73]

135. Secondary Outcome: Change From Baseline in Number of Steps Per Day (Week 16)
Description: Change from baseline in number of steps per day (week 16)
Time Frame: baseline, week 16
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 171 | 183
Steps | -655.04 (231.90) | -396.21 (217.31)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.318, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 258.83, 95% CI [-250.37 to 768.03]

136. Secondary Outcome: Change From Baseline in Number of Steps Per Day (Week 20)
Description: Change from baseline in number of steps per day (week 20)
Time Frame: baseline, week 20
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 172 | 182
Steps | -408.34 (247.32) | -197.17 (232.96)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.450, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 211.18, 95% CI [-338.04 to 760.39]

137. Secondary Outcome: Change From Baseline in Number of Steps Per Day (Week 24)
Description: Change from baseline in number of steps per day (week 24)
Time Frame: baseline, week 24
Population: as for outcome 103
Measure: Least Squares Mean (Standard Error); unit: Steps
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 167 | 186
Steps | -234.80 (261.49) | -183.34 (232.69)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; tiotropium versus placebo; Test type: Superiority or Other; p = 0.858, ANCOVA — [p-value comment as in outcome 5, analysis 1]; terms for treatment, site, and baseline value Mean Difference (Final Values) means difference in LSMeans; Mean Difference (Final Values) = 51.46, 95% CI [-512.20 to 615.12]

ADVERSE EVENTS:
Time Frame: First drug administration until 30 days after last drug administration
Arm/Group | Placebo | Tiotropium
Serious Adverse Events (participants affected / at risk) | 11/219 | 10/238
Other Adverse Events (participants affected / at risk) | 31/219 | 26/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=219) | Tiotropium (N=238)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=219) | Tiotropium (N=238)
Nasophayngitis (Infections and infestations) | 11 | 16
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 | 11

LIMITATIONS AND CAVEATS:
For individual outcome measures, only timepoints that had data collected are presented here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.